CLINICAL TRIAL: NCT04703855
Title: Post Market Surveillance of the HeartMate 3 Left Ventricular Assist System in Hong Kong and Taiwan
Brief Title: Hong Kong and Taiwan HM3 PMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment and regulatory status change
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10382; CRD 1022 (Other: Other Study ID Number)
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Advanced Heart Failure
Keywords: HeartMate 3; Left ventricular assist device; ABT-CIP-10382

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HeartMate 3™ left ventricular assist system (HM3 LVAS) (Experimental): Patients will be implanted with the HM3 LVAS
  Interventions: Device: HeartMate 3™ left ventricular assist system (HM3 LVAS)

INTERVENTIONS:
Device: HeartMate 3™ left ventricular assist system (HM3 LVAS) — Advanced heart failure patients will be implanted with the HM3 LVAS

SUMMARY:
Hong Kong and Taiwan HM3 PMS is a prospective, single arm, post market surveillance is designed to evaluate clinical and functional outcomes with the HM3 LVAS as a treatment for advanced heart failure. The PMS will enroll approximately 30 patients, that meet the HM3 commercially approved labelling indications, from approximately 4 sites in Hong Kong and Taiwan. PMS participants will be followed until the 24 months follow-up visit or until they experience an outcome, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

- All patients at the participating sites that are determined to meet the HM3 commercially approved labelling indication and have a planned HM3 implant are eligible to participate in this PMS. Assessment for eligibility criteria is based on medical records of the site and interview with a candidate patient.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gazzola, B. Sc., Study Director — Abbott Medical Devices
Locations (3):
- University of Hong Kong, Hong Kong, Pokfulam, Hong Kong
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Heart Transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 47.3 [29 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
NYHA [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity.Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients
  Participants
    Class IV | 3
    Class IIIB | 0
    Class IIIA | 0
    Class II | 0
    Class I | 0
INTERMACS [Count of Participants; unit: Participants] — INTERMACS Profiles describe the Heart Failure stage of the patients
  1. Critical cardiogenic shock
  2. Progressive decline on inotropic support
  3. Stable but inotrope dependent
  4. Resting symptoms home on oral therapy
  5. Exertion intolerant
  6. Exertion limited
  7. Advanced NYHA Class III symptom
  Participants
    1 | 0
    2 | 1
    3 | 2
    4 | 0
    5 | 0
    6 | 0
    7 | 0
Indication [Count of Participants; unit: Participants]
  Bridge to Transplant | 3
  Destination Therapy | 0
  Other Indications | 0
LVEF [Mean (Full Range); unit: percentage of LVEF] | 17.3 [10 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Number of Participants With Overall Survival to Transplant, Myocardial Recovery or on Device Support Free of Debilitating Stroke (Modified Rankin Score >3) or Reoperation for Pump Replacement
Description: Overall survival to transplant, myocardial recovery or on device support free of debilitating stroke (Modified Rankin Score >3) or reoperation for pump replacement will be assessed using the Kaplan-Meier product-limit method along with a competing outcomes graph. Subjects who are urgently transplanted due to a HeartMate 3 malfunction will be considered to have experienced a primary endpoint event, as will subjects who expire, suffer a debilitating stroke or have their HeartMate 3 exchanged due to a device failure. Subjects who are transplanted (except as described above), explanted for recovery, withdraw from the trial or are lost to follow-up will be censored at that time in the analysis.
Time Frame: Up to 6 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Primary Safety Endpoint: Number of Cumulative Occurrence of Adverse Events
Description: Cumulative occurrence of adverse events will be presented as percent of patients with adverse events
Time Frame: Up to 6 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Mean Change in Six-minute Walk Test From Baseline
Description: The 6-minute Walk test will be conducted at all follow-up visits until the end of the surveillance period.
Time Frame: Baseline and 1 Month post-implant
Population: Three subjects performed the assessment at Baseline and 1-Month, while two performed at 3 Months and one at 6 months (study premature end)
Measure: Mean (Standard Deviation); unit: meters
Groups:
- HeartMate 3™ Left Ventricular Assist System (HM3 LVAS): Patients implanted with the HeartMate 3™ left ventricular assist system (HM3 LVAS)
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
meters
  Baseline | 175.3 (159.0)
  1 Month post-implant | 197.3 (248.2)

4. Secondary Outcome: Change Proportion of New York Heart Association (NYHA) Functional Status From Baseline
Description: Subjects' NYHA Functional Status will be assessed at all scheduled follow-up visits until the end of the surveillance period.
  The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: Baseline and 1 Month post-implant
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
Unit on a scale
  Baseline | 4 (0)
  1-Month follow-up | 2 (1)

5. Secondary Outcome: Mean Change in EQ-5D-5L VAS Quality of Life (QoL) From Baseline
Description: The subject's quality of life will be measured by the EQ-5D-5L QoL questionnaire at baseline and all visits after the HM3 implant until the end of the surveillance period.
  EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Time Frame: Baseline and 1 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
score on a scale
  Baseline | 63.3 (12.6)
  1 Month post-implant | 83.3 (15.3)

6. Secondary Outcome: Frequency of Rehospitalization and Reoperation
Description: Frequency and reason will be reported for rehospitalization and reoperation.
Time Frame: Up to 6 months follow-up
Measure: Number; unit: number of events
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
number of events
  Rehospitalizations | 1
  Reoperations | 2

7. Secondary Outcome: Number of Participants With Device Malfunctions
Description: All suspected HM3 device malfunctions will be reported.
Time Frame: Up to 6 months follow-up
Measure: Number; unit: number of patients
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
Number analyzed (Participants) | 3
number of patients | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until study early termination. One subjects was followed until 6 months follow-up, while two reached 3 months visits
Arm/Group | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS) (N=3)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate 3™ Left Ventricular Assist System (HM3 LVAS) (N=3)
Cardiac Arrhythmias (Cardiac disorders) | 1 (2)
Neurological dysfunctions (Nervous system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The trial has been prematurely ended. Three 3 subjects were enrolled of which 2 have reached their 3 months follow-up and 1 reached 6 months at the time of study interruption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04703855/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04703855/SAP_001.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04703855/ICF_003.pdf